CLINICAL TRIAL: NCT03270072
Title: The Differential Impact of Proton Beam Irradiation Versus Conventional Radiation on Organs-at-risk in Stage II-III Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Beth Jimenez, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 17-031
Record Dates: First submitted 2017-06-13; First posted 2017-09-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Photon Therapy: The patients being treated on the Radiotherapy Comparative Effectiveness (RADCOMP) Consortium Trial (NCT02603341) at Massachusetts General Hospital that were randomized to receive photon therapy.
- Proton Therapy: The patients being treated on the Radiotherapy Comparative Effectiveness (RADCOMP) Consortium Trial (NCT02603341) at Massachusetts General Hospital that were randomized to receive proton therapy

SUMMARY:
The objective of the study is to serve as a correlative study for patients enrolled on the RadCOMP trial (NCT02603341), a randomized phase III study of stage II and III breast cancer patients treated with either conventional photon radiation or proton beam radiation

ELIGIBILITY:
Inclusion Criteria:

* Eligible for and scheduled to receive radiation therapy on Radiation Therapy Oncology Group (RTOG) Trial 3510 (Pragmatic Phase III Randomized Trial of Proton vs Photon Therapy for Patients with Non-Metastatic Breast Cancer Receiving Comprehensive Nodal Radiation: A Radiotherapy Comparative Effectiveness (RADCOMP) Consortium Trial). (NCT02603341)
* Ability to understand and the willingness to sign a study-specific written informed consent document

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled at Massachusetts General Hospital on the Radiation Therapy Oncology Group (RTOG) Trial 3510 (Pragmatic Phase III Randomized Trial of Proton vs Photon Therapy for Patients with Non-Metastatic Breast Cancer Receiving Comprehensive Nodal Radiation: A Radiotherapy Comparative Effectiveness (RADCOMP) Consortium Trial). (NCT02603341).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Global Longitudinal Strain (GLS) | Baseline, 6 Months
  Comparison of the change in GLS between conventional radiation and proton beam radiation groups. Participants who decrease their GLS by at least 2% 6-8 months following radiation therapy will be considered to demonstrate a significant decrement in GLS.

SECONDARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) Using Echocardiography | Baseline, end of treatment (approximately 10 weeks), then 6, 12, 24, 36, and 60 months post treatment
  Comparison of the change in LVEF between conventional radiation and proton beam radiation groups. Reduced cardiac function is defined as an ejection fraction <50%.
Radiation-induced Lung Parenchymal Changes Using CT Imaging | Baseline, 3,6,12, months post treatment
  Radiation-induced lung parenchymal changes will be assess with non-contrast enhanced computerized tomography (CT) scans and incidence will be estimated in each radiation group by the cumulative incidence function and compared using Gray's test. Among patients who do not have any changes detected, death and disease progression will be considered as competing risks.
Incidence of Thyroid Dysfunction | Baseline, end of treatment (approximately 10 weeks), then 12, 24, 36, and 60 months post treatment
  Incidence of thyroid insufficiency will be estimated in each radiation group by the cumulative incidence function and compared using Gray's test. In the absence of thyroid dysfunction, death and disease progression will be considered as competing risks.
Incidence of Ipsilateral Arm Lymphedema | Baseline, end of treatment (approximately 10 weeks), then 6, 12, 24, 36, and 60 months post treatment
  Incidence of ipsilateral arm lymphedema will be estimated in each radiation group by the cumulative incidence function and compared using Gray's test.
Severity of Ipsilateral Arm Lymphedema | Baseline, end of treatment (approximately 10 weeks), then 6, 12, 24, 36, and 60 months post treatment
  Serial arm measurements may be analyzed using mixed effects model to compare the severity of ipsilateral arm lymphedema over time between the radiation groups.
Ipsilateral Breast/Chest Wall Cosmesis | Baseline, end of treatment (approximately 10 weeks), then 6, 12, 24, 36, and 60 months post treatment
  Breast cosmesis will be assessed with characteristics graded on a four-point scale. Assessments will be performed by a trained nurse/nurse practitioner using the European Organization for Research and Treatment of Cancer (EORTC) Cosmetic Rating System for Breast Cancer. Incidence of adverse cosmesis (2=fair or 3=poor score) will be estimated in each radiation group by the cumulative incidence function and compared using Gray's test. Among patients without adverse breast cosmesis, death and disease progression will be considered as competing risks.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jimenez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States